CLINICAL TRIAL: NCT01071096
Title: Calcitonin Gene-related Peptide (CGRP) Levels in the Pathogenesis of Chronic Migraine
Brief Title: Calcitonin Gene-related Peptide Levels in Chronic Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cady, Roger, M.D. (Individual)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10-001AL
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Results first posted 2012-02-17 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Migraine
Keywords: Botox; OnabotulinumtoxinA; Chronic Migraine; Calcitonin Gene-Related Peptide; Saliva
MeSH Terms: interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OnabotulinumtoxinA (Active Comparator): Minimum dose of 155 international units (U) OnabotulinumtoxinA Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven specific head/neck muscle areas.
  Interventions: Drug: OnabotulinumtoxinA
- Saline (Placebo Comparator): 155 U Saline administered at 31 fixed-site, fixed-dose injections across seven specific head/neck muscle areas.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: OnabotulinumtoxinA — Minimum dose of 155 U OnabotulinumtoxinA Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven specific head/neck muscle areas. Subjects will continue to monitor headache symptoms with a headache diary and collect saliva samples as instructed.
  At investigator's discretion, additional 40 U OnabotulinumtoxinA Purified Neurotoxin Complex may be administered unilaterally or bilaterally, using follow-the-pain paradigm.
  Other Names: Botulinum Toxin Type A Purified Neurotoxin Complex; Botox
  Arms: OnabotulinumtoxinA
Drug: Saline — 155 U Saline administered at 31 fixed-site, fixed-dose injections across seven specific head/neck muscle areas. Subjects will continue to monitor headache using a headache diary and collect saliva samples as instructed.
  At investigator's discretion, additional Saline may be administered unilaterally or bilaterally, using follow-the-pain paradigm.
  Other Names: Placebo
  Arms: Saline

SUMMARY:
Twenty patients will be enrolled in a 2-site, 7-month, double-blind study conducted to evaluate a reduction in headache days and attacks and calcitonin gene-related peptide (CGRP) levels in saliva following treatment with OnabotulinumtoxinA versus saline.

Eligible patients will be randomized and receive injections of OnabotulinumtoxinA or Saline at Visit 1. Following 3 months plus a 1 month wash out, patients will receive cross-over injections at Visit 5.

Patients will return for monthly visits and exit the study at Visit 8.

Patients will collect saliva at monthly intervals and document in a daily headache diary throughout the study .

DETAILED DESCRIPTION:
This double-blind study will evaluate reduction in number of headache days following treatment with OnabotulinumtoxinA versus Saline. Additionally, CGRP levels in saliva will be correlated with a reduction in headache attacks.

At Visit 1, eligible subjects will be randomized 1:1 to receive injections of OnabotulinumtoxinA or Saline in an identical manner. Subjects will collect 3 saliva samples during each month of the 7 month study: 1 collection at Baseline headache level, 1 collection at onset of headache that is one degree worse than Baseline level that will be treated with acute therapy, and 1 collection at 2 hours following treatment. Subjects will document headache and headache symptoms in a daily diary and return to the clinic with diary and saliva samples at monthly visits.

Following 4 months (including a 1 month washout after Visit 4), subjects will return at Visit 5 and receive cross-over injections. Subjects randomized to OnabotulinumtoxinA at Visit 1 will receive injections of Saline. Subjects randomized to saline at Visit 1 will receive injections of OnabotulinumtoxinA. Subjects will document headache and headache symptoms in a daily diary and return to the clinic with diary and saliva samples at monthly visits.

At Visit 8, 3 months following re-injection at Visit 5, subjects will exit the study.

ELIGIBILITY:
Inclusion Criteria:

* must be outpatient, male or female, of any race, between 18 and 65 years of age.
* if female of childbearing potential must have negative pregnancy test result at Screening Visit and practice reliable method of contraception.

A female is considered of childbearing potential unless she is post menopausal for at least 12 months prior to administration of study drug, without a uterus and/or both ovaries or has been surgically sterilized for at least 6 months prior to study drug administration.

Reliable methods of contraception are: Complete abstinence from intercourse from 2 weeks prior to administration of the investigational product, throughout the study, and for a time interval (5 days) after completion or premature discontinuation from the study; or, History of bilateral tubal ligation; or, Sterilization of male partner; or, Implants of levonorgestrel; or, Injectable progestogen; or, Oral contraceptive (combination therapy with ethinyl estradiol plus a progestin) with a placebo week every 1-3 months; or, Any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per year (not all IUD's meet this criterion) in use at least 30 days prior to study drug administration; or, Spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a female diaphragm); or, Any other barrier methods (only is used in combination with any of the above acceptable methods) in use at least 14 days prior to study drug administration; or, Any other methods with published data showing that the highest expected failure rate for that methods is less than 1% per year.

* must have history of chronic migraine (with or without aura) according to the criteria proposed by the Headache Classification Committee of the International Headache Society (IHS) for at least 3 months prior to enrollment.
* must be able to understand the requirements of the study including maintaining a headache Diary, and signing informed consent.
* must be in good general health as determined by investigator.
* if taking migraine preventive, must be on a stable dose of preventive medication for at least 3 months prior to screening.

Exclusion Criteria:

* if female, is pregnant, planning to become pregnant during the study period, is breast feeding, or is of childbearing potential and not practicing a reliable form of birth control.
* has headache disorders outside IHS-defined chronic migraine definition.
* has evidence of underlying pathology contributing to their headaches.
* has any pathology of the salivary glands such as sialadenitis (e.g. Sjogren's syndrome, viral or bacterial sialadenitis) or condition or symptom that would alter the content of saliva.
* has any medical condition that may increase their risk with exposure to OnabotulinumtoxinA including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function.
* has profound atrophy or weakness of muscles in the target areas of injection.
* has skin conditions or infections at any of the injection sites.
* has allergy or sensitivities to any component of the test medication.
* who in the opinion of the investigator, has active major psychiatric or depressive disorders including alcohol/drug abuse.
* meets International Headache Society criteria for Medication Overuse with opioid or butalbital containing products.
* is planning or requiring surgery during the study.
* has a history of poor compliance with medical treatment.
* is currently participating in an investigational drug study or has participated in an investigational drug study within the previous 30 days of the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, MD, Principal Investigator — Clinvest
Locations (2):
- United States (2):
  - Clinvest, Springfield, Missouri
  - Island Neurological Associates, P.C., Plainview, New York

REFERENCES:
- [Background] Bellamy JL, Cady RK, Durham PL. Salivary levels of CGRP and VIP in rhinosinusitis and migraine patients. Headache. 2006 Jan;46(1):24-33. doi: 10.1111/j.1526-4610.2006.00294.x. PMID 16412148
- [Background] Cady RK, Vause CV, Ho TW, Bigal ME, Durham PL. Elevated saliva calcitonin gene-related peptide levels during acute migraine predict therapeutic response to rizatriptan. Headache. 2009 Oct;49(9):1258-66. doi: 10.1111/j.1526-4610.2009.01523.x. PMID 19788468
- [Background] Durham PL, Cady R, Cady R. Regulation of calcitonin gene-related peptide secretion from trigeminal nerve cells by botulinum toxin type A: implications for migraine therapy. Headache. 2004 Jan;44(1):35-42; discussion 42-3. doi: 10.1111/j.1526-4610.2004.04007.x. PMID 14979881
- [Background] Bruno PP, Carpino F, Carpino G, Zicari A. An overview on immune system and migraine. Eur Rev Med Pharmacol Sci. 2007 Jul-Aug;11(4):245-8. PMID 17876959
- [Background] Perini F, D'Andrea G, Galloni E, Pignatelli F, Billo G, Alba S, Bussone G, Toso V. Plasma cytokine levels in migraineurs and controls. Headache. 2005 Jul-Aug;45(7):926-31. doi: 10.1111/j.1526-4610.2005.05135.x. PMID 15985111
- [Background] Sarchielli P, Alberti A, Vaianella L, Pierguidi L, Floridi A, Mazzotta G, Floridi A, Gallai V. Chemokine levels in the jugular venous blood of migraine without aura patients during attacks. Headache. 2004 Nov-Dec;44(10):961-8. doi: 10.1111/j.1526-4610.2004.04189.x. PMID 15546258
- [Background] Munno I, Marinaro M, Bassi A, Cassiano MA, Causarano V, Centonze V. Immunological aspects in migraine: increase of IL-10 plasma levels during attack. Headache. 2001 Sep;41(8):764-7. doi: 10.1046/j.1526-4610.2001.01140.x. PMID 11576199

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Subjects were injected with OnabotulinumtoxinA at Visit 1 (Day 1) and followed for 3 months through monthly office visits (Visits 2, 3, and 4 at Days 31, 61 and 91). Subjects went through a 1 month (30 day) washout period between Visit 4 (Day 91) and Visit 5 (Day 121). Subjects were injected with Saline at Visit 5 (Day 121) and followed for 3 months through monthly office visits (Visits 5, 6, and 7 at Days 151, 181, and 211).
- Group B: Subjects were injected with Saline at Visit 1 (Day 1) and followed for 3 months through monthly office visits (Visits 2, 3, and 4 at Days 31, 61 and 91). Subjects went through a 1 month (30 day) washout period between Visit 4 (Day 91) and Visit 5 (Day 121). Subjects were injected with OnabotulinumtoxinA at Visit 5 (Day 121) and followed for 3 months through monthly office visits (Visits 5, 6, and 7 at Days 151, 181, and 211).
Period: First Intervention (90 Days)
Arm/Group | Group A | Group B
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Washout Period (30 Days)
Arm/Group | Group A | Group B
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0
Period: Second Intervention (90 Days)
Arm/Group | Group A | Group B
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Participants: Enrolled Participants includes subjects in both Group A (treated with BOTOX and Visit 1 and Placebo at Visit 5) and Group B (treated with Placebo at Visit 1 and BOTOX at Visit 5).
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48.45 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Headache Days Per Month From Baseline (BL) to Months 1 Through 7.
Description: Baseline number of headache days per month collected historically at screening. Post-treatment number of headache days collected per month via diary.
Time Frame: Baseline (collected historically at screening) versus (vs.) Month (Mo) 1, Mo 2, Mo 3, Mo 4, Mo 5, Mo 6, and Mo 7
Measure: Mean (Standard Deviation); unit: days
Groups:
- Group A: OnabotulinumtoxinA at Visit 1 (headache days in Months 1, 2 and 3) and Saline at Visit 5 (headache days in Months 5, 6 and 7) with washout and crossover at Month 4
- Group B: Saline at Visit 1 (headache days in Months 1, 2 and 3) and OnabotulinumtoxinA at Visit 5 (headache days in Months 5, 6 and 7) with washout and crossover at Month 4
Arm/Group | Group A | Group B
Number analyzed (Participants) | 9 | 10
days
  Baseline vs. Month 1 | -7.61 (8.01) | -6.67 (6.28)
  Baseline vs. Month 2 | -9.72 (5.96) | -5.22 (4.44)
  Baseline vs. Month 3 | -10.06 (5.92) | -5.22 (5.14)
  Baseline vs. Month 4 | -9.50 (8.34) | -6.89 (7.08)
  Baseline vs. Month 5 | -8.94 (8.15) | -6.33 (4.12)
  Baseline vs. Month 6 | -9.50 (7.93) | -9.22 (5.45)
  Baseline vs. Month 7 | -6.50 (7.53) | -4.56 (6.89)

2. Primary Outcome: Change in Number of Headache Days Per Month From Baseline to Month 1 (M1), Month 1 to Month 2 (M2), and Month 2 to Month 3 (M3).
Description: as for outcome 1
Time Frame: Baseline (collected historically at screening) vs. Mo 1, Mo 1 vs. Mo 2, Mo 2 vs. Mo 3, Mo 3 vs. Mo 4, Mo 4 vs. Mo 5, Mo 5 vs. Mo 6, and Mo 6 vs. Mo 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 9 | 10
days
  Baseline vs. Mo 1 | -7.61 (8.01) | -6.67 (6.28)
  Mo 1 vs. Mo 2 | -2.11 (7.20) | 1.44 (7.78)
  Mo 2 vs. Mo 3 | -0.33 (3.97) | 0.00 (1.94)
  Mo 3 vs. Mo 4 | 0.56 (3.91) | -1.67 (5.66)
  Mo 4 vs. Mo 5 | 0.56 (3.21) | 0.56 (4.61)
  Mo 5 vs. Mo 6 | -0.56 (3.84) | -2.89 (5.42)
  Mo 6 vs. M 7 | 3.00 (3.84) | 4.67 (5.63)

3. Secondary Outcome: Inter-ictal (Baseline) Levels of Saliva Calcitonin Gene-related Peptide (CGRP)
Description: CGRP Level collected each month when subject did not have a headache or was at lowest pain level of headache that month.
Time Frame: Baseline levels collected for OnabotulinumtoxinA and Saline treatment during Months 1 through 7
Measure: Mean (Standard Error); unit: pmol/mg total protein
Groups:
- OnabotulinumtoxinA: This group is a combination of information gathered from both groups while treating with OnabotulinumtoxinA: Group A (Months 1-3) and Group B (Months 5-7).
- Saline: This group is a combination of information gathered from both groups while treating with Saline: Group A (Months 5-7) and Group B (Months 1-3).
Arm/Group | OnabotulinumtoxinA | Saline
Number analyzed (Participants) | 19 | 19
pmol/mg total protein
  Treatment Month 1 | 39.64 (7.5) | 40.79 (9.73)
  Treatment Month 2 | 28.37 (7.07) | 39.14 (9.74)
  Treatment Month 3 | 26.14 (3.93) | 50.63 (15.04)

4. Secondary Outcome: Saliva CGRP Levels for OnabotulinumtoxinA Responders (Reduction of Headache Days Greater Than 30%) vs. Non-responders and Saline
Description: Saliva samples collected at Baseline (at no headache or lowest level of headache), at headache attack directly before taking rescue medication and 2 hours after treating with rescue medication.
Time Frame: For OnabotulinumtoxinA and Saline treatment months 1, 2 and 3
Measure: Mean (Standard Deviation); unit: pmol/mg total protein
Groups:
- OnabotulinumtoxinA Responders: This group is a combination of information gathered from both groups while treating with OnabotulinumtoxinA: Group A (Months 1-3) and Group B (Months 5-7). Includes subjects with >30% reduction in number of headache days per month when compared to Baseline
- OnabotulinumtoxinA Non-Responders: This group is a combination of information gathered from both groups while treating with OnabotulinumtoxinA: Group A (Months 1-3) and Group B (Months 5-7). Includes subjects with <30% reduction in number of headache days per month when compared to Baseline
Arm/Group | OnabotulinumtoxinA Responders | OnabotulinumtoxinA Non-Responders | Saline
Number analyzed (Participants) | 10 | 9 | 19
pmol/mg total protein
  Treatment Month 1 - Baseline | 52.36 (56.31) | 29.36 (32.81) | 70.46 (98.26)
  Treatment Month 1 - Attack | 27.94 (21.85) | 22.36 (20.38) | 36.23 (33.16)
  Treatment Month 1 - 2 Hours Post | 61.55 (44.82) | 23.66 (12.11) | 39.76 (54.51)
  Treatment Month 2 - Baseline | 59.89 (49.27) | 28.66 (20.59) | 44.12 (49.70)
  Treatment Month 2 - Attack | 60.14 (51.18) | 32.65 (33.80) | 33.05 (30.96)
  Treatment Month 2 - 2 Hours Post | 39.13 (60.98) | 22.35 (19.94) | 33.93 (35.91)
  Treatment Month 3 - Baseline | 51.33 (77.44) | 32.61 (40.13) | 58.74 (53.86)
  Treatment Month 3 - Attack | 73.18 (58.88) | 30.17 (38.63) | 46.16 (40.29)
  Treatment Month 3 - 2 Hours Post | 54.04 (34.77) | 19.11 (13.24) | 49.39 (43.81)

5. Secondary Outcome: Changes Between Inter-ictal (Baseline) Levels Between Responders and Non-responders
Description: Only cytokines with a mean densimetric value 1.65 times the background grey value in a minimum of 3 patients were considered detectable. These are reported below. Values normalized to positive control array spots after background subtraction: C5/C5a, CD40 Ligand, Granulocyte Colony Stimulating Factor (G-CSF), Growth Regulated Oncogene(GRO)-alpha, Soluble Intercellular Adhesion Molecule (sICAM)-1, Interferon gamma (IFN-y), Interleukin(IL)-1alpha, 1beta, 1ra, 8, 16, 17E, & 23, Interferon Gamma-Induced Protein 10 (IP-10), Interferon-inducible T cell alpha chemoattractant (I-TAC), Macrophage Migration Inhibitory Factor (MIF), Serpin E1, and Regulated Upon Activation Normal T-cell Expressed (RANTES)
Time Frame: For OnabotulinumtoxinA and Saline treatment months 1, 2 and 3 at Baseline level (inter-ictal) and at onset of headache that is one degree worse than Baseline level and that will be treated with acute therapy
Population: Number of Participants Analyzed is low due to some unusable samples and missing samples making comparison between months impossible. 5 Responders and 5 Non-Responders provided enough samples at all time points for comparisons.
Measure: Mean (Standard Deviation); unit: Florescent Units (FU)
Groups:
- Month 1 vs. Saline Responders: Fold change between first treatment months with OnabotulinumtoxinA and Saline in subjects with >30% reduction in number of headache days per month from baseline.
- Month 1 vs. Saline Non-Responders: Fold change between first treatment months with OnabotulinumtoxinA and Saline in subjects with <30% reduction in number of headache days per month from baseline.
- Month 3 vs. Saline Responders: Fold change between third treatment months with OnabotulinumtoxinA and Saline in subjects with >30% reduction in number of headache days per month from baseline.
- Month 3 vs. Saline Non-Responders: Fold change between third treatment months with OnabotulinumtoxinA and Saline in subjects with <30% reduction in number of headache days per month from baseline.
- Month 1 vs. Month 3 Responders: Fold change between first and third treatment months with OnabotulinumtoxinA in subjects with >30% reduction in number of headache days per month from baseline.
- Month 1 vs. Month 3 Non-Responders: Fold change between first and third treatment months with OnabotulinumtoxinA in subjects with <30% reduction in number of headache days per month from baseline.
Arm/Group | Month 1 vs. Saline Responders | Month 1 vs. Saline Non-Responders | Month 3 vs. Saline Responders | Month 3 vs. Saline Non-Responders | Month 1 vs. Month 3 Responders | Month 1 vs. Month 3 Non-Responders
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
Florescent Units (FU)
  C5/C5a | 1.38 (0.23) | 1.01 (0.90) | 1.39 (0.80) | 1.61 (0.54) | 1.03 (0.57) | 3.26 (3.35)
  CD40 Ligand | 1.09 (0.25) | 1.26 (0.99) | 0.98 (0.37) | 1.31 (0.63) | 0.91 (0.27) | 1.22 (0.40)
  G-CSF | 0.92 (0.45) | 0.93 (0.55) | 0.85 (0.24) | 0.99 (0.58) | 1.07 (0.74) | 1.34 (0.76)
  GROa | 1.34 (1.56) | 3.18 (2.20) | 1.40 (1.33) | 1.81 (1.32) | 1.05 (0.96) | 0.73 (0.55)
  sICAM-1 | 2.60 (2.32) | 0.61 (0.54) | 5.99 (6.13) | 2.00 (1.98) | 3.99 (3.22) | 1.51 (0.15)
  IFN-y | 1.29 (0.34) | 0.80 (0.69) | 1.29 (0.82) | 1.92 (2.95) | 0.91 (0.34) | 1.63 (0.94)
  IL-1alpha | 2.30 (1.86) | 2.88 (4.29) | 1.50 (0.92) | 2.14 (3.04) | 0.86 (0.60) | 0.81 (0.32)
  IL-1beta | 1.63 (0.80) | 1.12 (1.09) | 1.38 (1.15) | 0.51 (0.23) | 1.15 (0.12) | 1.03 (0.43)
  IL-1ra | 1.13 (0.56) | 2.02 (2.66) | 0.96 (0.39) | 1.90 (1.58) | 0.88 (0.12) | 1.30 (0.43)
  IL-8 | 1.61 (0.83) | 1.70 (2.03) | 2.71 (2.29) | 1.22 (1.24) | 4.38 (6.98) | 2.28 (NA) — Only one value available (2.28) so there is no standard deviation between reported values.
  IL-16 | 0.91 (0.63) | 2.07 (1.63) | 0.75 (0.48) | 1.97 (1.64) | 0.98 (0.66) | 1.10 (0.48)
  IL-17E | 0.86 (0.50) | 1.02 (0.91) | 1.59 (1.79) | 0.42 (0.13) | 1.28 (0.85) | 1.45 (0.04)
  IL-23 | 2.45 (1.85) | 1.80 (1.55) | 1.06 (0.12) | 1.69 (1.54) | 0.93 (0.01) | 2.61 (3.34)
  IP-10 | 1.32 (1.05) | 0.95 (0.17) | 0.86 (0.52) | 2.76 (2.23) | 1.55 (1.50) | 3.11 (2.69)
  I-TAC | 1.40 (0.78) | 0.28 (0.12) | 1.01 (0.89) | 0.94 (0.26) | 0.67 (0.27) | 3.65 (1.33)
  MIF | 3.71 (6.25) | 9.55 (19.47) | 2.71 (4.50) | 8.66 (16.79) | 0.80 (0.32) | 1.24 (0.27)
  Serpin E1 | 0.98 (0.17) | 0.70 (0.53) | 0.70 (0.33) | 0.90 (0.82) | 0.76 (0.39) | 3.16 (3.25)
  RANTES | 0.95 (0.41) | 0.77 (0.28) | 0.93 (0.41) | 0.91 (0.27) | 1.14 (0.21) | 1.24 (0.26)

ADVERSE EVENTS:
Groups:
- Saline: Subjects injected with Saline in Group A at Visit 5 (Day 151) and Group B at Visit 1 (Day 1)
- OnabotulinumtoxinA: Subjects injected with onabotulinumtoxinA in Group A at Visit 1 (Day 1) and Group B at Visit 5 (Day 151)
Arm/Group | Saline | OnabotulinumtoxinA
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 11/20 | 15/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline (N=20) | OnabotulinumtoxinA (N=20)
1st Degree Burn on Extremity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
2nd Degree Burn on Extremity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Contusion of extremity (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dental Implant (Surgical and medical procedures) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated Cholesterol (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Enlarged Lymph Node (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Eyebrow Ptosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Facial Edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fibromyalgia Pain (Nervous system disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Head Pain (General disorders) | 0 (0) | 1 (1)
Head Tenderness (General disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Heart Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Herpes Zoster (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hoarseness (General disorders) | 1 (1) | 0 (0)
Influenza (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inner Ear Fluid Imbalance (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Oral Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Otitis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Paresthesia as Injection Site (Nervous system disorders) | 0 (0) | 1 (1)
Parotid Glad Infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngitis Streptococcal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Respiratory Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ruptured Breast Implant (Surgical and medical procedures) | 0 (0) | 1 (1)
Salivary Gland Infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary Gland Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Scalp Pain (General disorders) | 0 (0) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Stress (General disorders) | 0 (0) | 1 (1)
Upper Respiratory Track Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Vertigo (General disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to identified lab errors related to processing of samples for CGRP and cytokine levels, samples are currently being re-processed. Results will be posted following re-analysis of all study data related to sample values.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No